CLINICAL TRIAL: NCT02584400
Title: Non-invasive Imaging of Tumor Hypoxia With [18F]HX4 Positron-Emission-Tomography (PET): A Phase II Trial
Brief Title: Tumor Hypoxia With HX4 PET in Several Diseases
Acronym: HX4 SD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: patients did not want to participate
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL50833.068
Record Dates: First submitted 2015-10-07; First posted 2015-10-22 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Prostatic Neoplasms; Esophageal Neoplasms; Neoplasm Metastases, Brain; Rectal Neoplasms; Brain Neoplasm, Primary
Keywords: prostatic tumors; [18F]HX4 Pet imaging; hypoxia; phase II trial; esophageal tumors; rectal tumors; brain metastases; primary brain tumors
MeSH Terms: conditions — Prostatic Neoplasms; Esophageal Neoplasms; Neoplasm Metastasis; Rectal Neoplasms; Brain Neoplasms; Hypoxia | interventions — Injections; 3-fluoro-2-(4-((2-nitro-1H-imidazol-1-yl)methyl)-1H-1,2,3-triazol-1-yl)propan-1-ol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [18F]HX4 PET imaging (Experimental): Injection with the hypoxia tracer [18F]HX4 and PET imaging at baseline for esophageal, rectal, prostate cancer, primary brain tumor (grade IV glioma) and brain metastases and after 2 weeks of radiotherapy for esophageal, rectal and brain metastases
  Interventions: Drug: Injection with the hypoxia tracer [18F]HX4,

INTERVENTIONS:
Drug: Injection with the hypoxia tracer [18F]HX4, — The [18F]HX4 PET scan will be performed, by administrating 444 MBq (12 mCi) [18F]HX4 via a bolus IV injection.
  Other Names: [18F]HX4 is 3-[18F]fluoro-2-(4-((2-nitro-1H-imidazol-1-yl)methyl)-1H-1,2,3-triazol-1-yl)propan-1-ol

SUMMARY:
Regulation of tissue oxygen homeostasis is critical for cell function, proliferation and survival. Evidence for this continues to accumulate along with our understanding of the complex oxygen-sensing pathways present within cells. Several pathophysiological disorders are associated with a loss in oxygen homeostasis, including heart disease, stroke, and cancer. The microenvironment of tumors in particular is very oxygen heterogeneous, with hypoxic areas which may explain our difficulty treating cancer effectively. Prostate carcinomas are known to be hypoxic. Increasing levels of hypoxia within prostatic tissue is related to increasing clinical stage, patient age and a more aggressive prostate cancer. Several researches indicated that hypoxia might also play a role in esophageal cancer. In glial brain tumors, hypoxia is correlated with more rapid tumor recurrence and the hypoxic burden in newly diagnosed glioblastomas is linked to the biological aggressiveness. In brain metastases CA-IX expression (a marker for hypoxia) is correlated to the primary non-small cell lung carcinomas. Hypoxia enhances proliferation, angiogenesis, metastasis, chemoresistance and radioresistance of hepatocellular carcinoma. The hypoxic markers HIF-1α, VEGF, CA-IX and GLUT-1 were all over expressed in colorectal cancer and its liver metastases. Based on literature, hypoxia in tumors originating or disseminated to prostate, esophagus, brain and rectum cancer will be studied in this trial.

DETAILED DESCRIPTION:
Rationale: Non-invasive imaging of hypoxia with the aid of PET-scans could help to select the patients having a hypoxic tumor, who could be treated with specific anti-hypoxic treatments. The added value of additional anti-hypoxic treatments depends on the presence of hypoxia and adequate patient selection. Several 2-nitroimidazoles, labeled with Fluor-18 (18F) have already been used in patients to identify hypoxia. However, suboptimal image quality and unpredictable kinetics limit their use. In extensive pre-clinical models and clinical trials the combination of HX4 labeled with 18F showed to be a promising and non-toxic new probe to determine hypoxia. With this tracer the proportion of hypoxic tumors in several cancer types will be verified.

Objective: Determine if tumor hypoxia can be accurately visualized with [18F]HX4 in solid lesions.

Study design: Phase II, several solid tumors, single-centre, imaging, non-randomized, open label trial.

Study population:

Main patient characteristics are:

* Histological/cytological confirmed carcinoma of de esophagus, rectum or prostate or radiological suspicion for Grade IV glioma (primary brain tumor) or brain metastases.
* WHO performance status 0 to 2
* Adequate renal function (calculated creatinine clearance at least 60 ml/min).
* Capable of complying with study procedures

Main intervention: In addition to standard clinical care patients receive two additional PET scans after injection with the hypoxia tracer [18F]HX4.

Main study parameters/endpoints:

* Visualization and quantification of tumor hypoxia with [18F] HX4 PET imaging
* Exploring the potential relationship between [18F] HX4 uptake with local and locoregional tumor recurrence and survival
* Correlation of hypoxia imaging with blood hypoxia markers
* Correlation of hypoxia imaging with tumor tissue biomarkers
* Evaluation of tumor hypoxia changes during treatment.
* Spatial correlation of [18F] HX4-PET with imaging pre-treatment (if present from routine clinical practice)
* Spatial correlation of [18F] HX4-PET with imaging three months after treatment (if present from routine clinical practice)
* Quantitative and qualitative correlation of [18F] HX4-PET obtained before treatment and two weeks into treatment

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The radiation burden due to [18F]HX4 is similar to that encountered in many routine nuclear medicine procedures e.g. [18F]FDG PET. Administration of [18F]HX4 presents no known risks. In previous studies (healthy volunteers, phase I, phase II) no adverse effects were observed. There are no immediate potential benefits except the satisfaction to participate to improve of knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytological confirmed carcinoma of de esophagus, rectum or prostate or radiological suspicion for Grade IV glioma (primary brain tumor) or brain metastases
* WHO performance status 0 to 2.
* Adequate renal function (calculated creatinine clearance at least 60 ml/min).
* The patient is willing and capable to comply with study procedures
* 18 years or older
* Have given written informed consent before patient registration

Exclusion Criteria:

* Recent (< 3 months) myocardial infarction
* Pregnant or breast feeding and willing to take adequate contraceptive measures during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-05; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Visualization of tumor hypoxia with [18F] HX4 PET imaging, valuated by the measurement of a tumor-to-background (T/B) ratio on the [18F]HX4 PET/CT | 4 years
  Visualization of tumor hypoxia with [18F] HX4 PET imaging
Quantification of tumor hypoxia with [18F] HX4 PET imaging, evaluated by the measurement of a tumor-to-background (T/B) ratio on the [18F]HX4 PET/CT | 4 years
  Quantification of tumor hypoxia with [18F] HX4 PET imaging

SECONDARY OUTCOMES:
Time between [18F] HX4 uptake with local and locoregional tumor recurrence and survival | 4 years
  Exploring the potential relationship of [18F] HX4 uptake with local and locoregional tumor recurrence and survival
Correlation of hypoxia imaging with blood hypoxia markers will be measured by the Pearson or Spearman correlation coefficient | 4 years
  Correlation of hypoxia imaging with blood hypoxia markers
Correlation of hypoxia imaging with tumor tissue biomarkers will be measured by the Pearson or Spearman correlation coefficient | 4 years
  Correlation of hypoxia imaging with tumor tissue biomarkers
Evaluation of tumor hypoxia changes during treatment by comparison of the PET uptake values in the tumor, measured before and during treatment | 4 years
  Evaluation of tumor hypoxia changes during treatment
Spatial correlation of [18F] HX4-PET with imaging pre-treatment using a correlation coefficient | 4 years
  Spatial correlation of [18F] HX4-PET with imaging pre-treatment (if present from routine clinical practice); performed by a rigid registration of the scans and a voxel wise comparison of the uptake within the tumor
Spatial correlation of [18F] HX4-PET with imaging three months after treatment using a correlation coefficient | 3 months
  Spatial correlation of [18F] HX4-PET with imaging three months after treatment (if present from routine clinical practice), performed by a rigid registration of the scans and a voxel wise comparison of the uptake within the tumor

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, Prof. dr., Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- MAASTRO Clinic, Maastricht, Limburg, Netherlands